CLINICAL TRIAL: NCT06254482
Title: A Phase 2b, Double-Blind, Randomized Extension Study to Evaluate the Long-Term Safety and Efficacy of Votoplam in Participants With Huntington's Disease
Brief Title: An Extension Study to Evaluate the Long-Term Safety and Efficacy of Votoplam in Participants With Huntington's Disease (HD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTC518-CNS-004-HD; 2023-504628-24-00 (Other: EU CT Number); CHTT227A12201 (Other: Novartis)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Huntington Disease
Keywords: Neurodegenerative disorder; Rare disease
MeSH Terms: conditions — Huntington Disease; Neurodegenerative Diseases; Rare Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Votoplam 5 mg (Experimental): Participants will receive Votoplam 5 mg tablets once daily orally for 48 months.
  Interventions: Drug: Votoplam
- Votoplam 10 mg (Experimental): Participants will receive votoplam 10 mg tablets once daily orally for 48 months.
  Interventions: Drug: Votoplam

INTERVENTIONS:
Drug: Votoplam — Votoplam will be administered per dose and schedule specified in the arm.
  Other Names: HTT227 / PTC518

SUMMARY:
The primary goal of this study is to evaluate the long-term safety and pharmacodynamic effects of votoplam in participants with HD.

DETAILED DESCRIPTION:
Participants who completed the Treatment Period in the parent Phase 2a Study PTC518-CNS-002-HD (NCT05358717), fulfilled the enrollment criteria, and chose to enroll in this extension study will undergo baseline evaluations and be assessed for 54 additional months.

All participants will receive active votoplam in this extension study. Participants who received votoplam in the parent Study PTC518-CNS-002-HD will continue at the same dose level they received in that study in a blinded fashion (5, 10 milligrams [mg]). Participants who received placebo in the parent Study PTC518-CNS-002-HD will be allocated to a votoplam dose level according to the same dosing group in which they were previously randomized (5, 10 mg).

ELIGIBILITY:
Inclusion Criteria:

* Participant who has completed the Treatment Period in Study PTC518-CNS-002-HD.

Exclusion Criteria:

* Participants who have not previously completed the Treatment Period in Study PTC518-CNS-002-HD.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2029-07-16 (Estimated); Study Completion 2029-07-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline up to Month 54
Blood Total Huntingtin Protein (tHTT) Levels | Baseline up to Month 52

SECONDARY OUTCOMES:
Change From Baseline in Caudate Volume as Assessed Via Volumetric Magnetic Resonance Imaging (vMRI) at Month 48 | Baseline, Month 48
Change From Baseline in Composite Unified Huntington's Disease Rating Scale (cUHDRS) Scores at Month 48 | Baseline, Month 48
Cerebrospinal Fluid (CSF) Mutant Huntingtin Protein (mHTT) Levels | Baseline up to Month 48
Blood mHTT Protein Levels | Baseline up to Month 52

CONTACTS AND LOCATIONS:
Locations (24):
- Australia (2):
  - Novartis Investigative Site, Clayton
  - Novartis Investigative Site, Westmead
- Novartis Investigative Site, Innsbruck, Austria
- Novartis Investigative Site, Ottawa, Canada
- France (3):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
- Italy (3):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, San Giovanni Rotondo
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Christchurch, New Zealand
- Spain (4):
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Madrid
- United Kingdom (4):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com